CLINICAL TRIAL: NCT06314308
Title: Community Health Worker Assisted Task Specific and Cognitive Therapy at Home With Exposure After Stroke
Acronym: CATCHES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Imama A. Naqvi, Assistant Professor of Neurology at the Columbia University Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAU8161; 5P30AG064198-05 (NIH)
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Stroke, Acute Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Task Specific Training Task-Specific Training (TST) which is the repeated, active practice of a motor skill or activity that is meaningful to an individual with the goal of skill acquisition and retention will be provided over 5 sessions after initial an initial assessment by a physical therapist. Cognitive Behavioral Therapy (CBT) with exposure is a psychotherapeutic intervention that focuses on modifying individuals' thoughts and behavior guided through graded exposure will be guided by a psychologist.
  Interventions: Behavioral: CATCHES

INTERVENTIONS:
Behavioral: CATCHES — At the baseline visit (T0), informed consent will be obtained, and baseline questionnaires and measurements completed. A physical activity monitor will be provided. After discharge, Task Specific Training guided by Cognitive Behavioral Therapy with Exposure delivered over 7 one-hour sessions including two intake sessions by specialists and five follow up sessions delivered by CHWs individually at home over 3 months. After the final session at 12 weeks (about 3 months), participants will complete a study end visit (T1) which will include follow up questionnaires and measurements.

SUMMARY:
CATCHES is a novel intervention for preliminary testing, integrating Task Specific Therapy at home guided by Community Health Workers (CHW) under supervision of a licensed Physical Therapist (PT) guided by telehealth based Cognitive Behavioral Therapy (CBT) to reduce task specific fears through repetitive exposure and adaptive behavioral activation strategies and facilitate engagement in physical activity.

1. To integrate and establish feasibility of CATCHES intervention. Hypothesis: A multidisciplinary team providing home based TST with exposure therapy tailored to an underserved urban setting will inform a patient-centered behavioral intervention to reduce fear of falling (FOF) among post-acute stroke patients returning home. Feasibility outcomes will include recruitment, retention, and fidelity of implementation.
2. Test effects of the intervention on hypothesized treatment mechanism of fear of falling. Hypothesis: Therapy will reduce task specific fear of falling Primary outcome will be change in Activities-specific Balance Confidence Scale.
3. Explore physical activity measures subjectively and objectively. Exploratory outcomes include pre and post Timed Up and Go test, patient reported outcome surveys and activity as measured by wearable devices.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability in the country, and ethno-racial inequities are persistent. Almost two thirds of stroke patients are discharged home without effective rehabilitation or community-based support. Falls can occur at home, and associated fear of falling leads to avoidance behaviors that limit physical activity and community reintegration. Here the investigators propose a novel intervention in a feasibility study for preliminary testing, integrating Task Specific Therapy at home guided by Community Health Workers (CHW) under supervision of a licensed Physical Therapist (PT) in conjunction with telehealth based Cognitive Behavioral Therapy (CBT) with reduce task specific fears through repetitive exposure and adaptive behavioral activation strategies to facilitate engagement in physical activity. The main objective is to assess the feasibility of this intervention. The secondary objective is to explore the underlying behavioral mechanism for behavior change and explore physical activity.

ELIGIBILITY:
Inclusion criteria:

* Aged over 18 years
* Plan for discharge home after stroke and ability to provide consent
* Low balance confidence (Activities-specific Balance Confidence < 80)

Exclusion criteria:

* Modified Rankin Scale > 2 at time of enrollment
* Severe Stroke (NIH Stroke Scale > 14 and/or significant aphasia, dysarthria, or cognitive impairment precluding ability to complete study questionnaires as determined by interviewer)
* Legal blindness precluding ability to view infographic or education materials
* Terminal non-cardiovascular illness (life expectancy < 1 year)
* Co-morbid mental illness requiring hospitalization
* Unavailable for follow-up
* Non-English and non-Spanish speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of intervention completers to demonstrate feasibility | 3 months
  This outcome is designed to measure intervention feasibility, which will take recruitment, retention, and fidelity of implementation into account. The participants who complete 100% of the study required procedures will be tallied.

SECONDARY OUTCOMES:
Change in Activities-specific Balance Confidence Scale Score | Baseline and 3 months
  This outcome is designed to measure the change in fear of falling. This is a 16-item self-reported questionnaire with a score range of 1-100. 1 = no confidence and 100 = completely confident. The higher the score, the lesser the fear. The scale score is calculated by dividing the total by 16.

OTHER OUTCOMES:
Timed Up and Go Test Score | Baseline, 3 months
  This exploratory outcome is to measure change in physical function. The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk in older adults. The test involves recording the length of time it takes a participant to stand from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. Change in time to perform the test will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Imama A Naqvi, MD, MS, Principal Investigator — Columbia University
Locations (1):
- The Neurological Institute of New York, Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No